CLINICAL TRIAL: NCT06888011
Title: Implementation of the New Pediatric Obesity Clinical Practice Guideline in Rural Families and Clinics: A Randomized Clinical Trial
Brief Title: iAmHealthy Clinical Practice Guideline (CPG)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00160797; R01NR021278 (NIH)
Record Dates: First submitted 2025-02-21; First posted 2025-03-21 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Obesity; Rural Health; Clinical Practice Guideline
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: The study is a multilevel factorial individually and cluster randomized stepped wedge design RCT with interventions targeted to the individual patient level (iAmHealthy vs. Newsletter) and to the clinic (Healthy Clinic).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Participants: iAmHealthy (Experimental): The iAmHealthy intervention is a rurally tailored empirically supported family-based behavioral group program targeting the families of children who are overweight or obese and providing 26 contact hours of group and individual intervention over six months.
  Interventions: Behavioral: Participants: iAmHealthy
- Participants: Newsletter (Active Comparator): Families will receive a monthly newsletter for six months.
  Interventions: Behavioral: Participants: Newsletter
- Clinics: Healthy Clinics (Other): Healthy Clinics is a clinic level intervention designed to improve provider office processes using a bundled intervention of provider prompts, skills training and intervention tools implemented with performance feedback. Clinics are randomized to the order in which they undertake the individually randomized iAmHealthy vs. Newsletter intervention and the cluster randomized Healthy Clinic intervention
  Interventions: Behavioral: Participants: iAmHealthy; Behavioral: Participants: Newsletter; Other: Clinics: Healthy Clinics

INTERVENTIONS:
Behavioral: Participants: iAmHealthy — Families will take part in an educational group program with parents and their children. These one-hour meetings will be focused on living healthy lifestyles and engaging in healthy habits as a family and will occur weekly for three months and monthly for three months. Each family will also have the opportunity to receive individual health coaching sessions every other week that will last approximately 30 minutes to address concerns and health behaviors specific to each pair. There will be additional opportunities to demonstrate and apply learned concepts.
  Arms: Clinics: Healthy Clinics; Participants: iAmHealthy
Behavioral: Participants: Newsletter — Families assigned to the newsletter control intervention will receive the AAP Healthy Children Newsletter (HealthyChildren.org) every month for six months.
  Arms: Clinics: Healthy Clinics; Participants: Newsletter
Other: Clinics: Healthy Clinics — Healthy Clinics is a clinic level intervention designed to improve provider office processes using a bundled intervention of provider prompts, skills training and intervention tools implemented with performance feedback. Each clinic receives Healthy Clinics at some point in the intervention.
  Arms: Clinics: Healthy Clinics

SUMMARY:
The current study is a multilevel factorial design RCT with interventions at the clinic (Healthy Clinic intervention period vs. Control period) and individual patient levels (iAmHealthy vs. Newsletter).

DETAILED DESCRIPTION:
Obesity poses a major health risk, contributing to elevated morbidity and mortality from cancer, cardiovascular disease, and diabetes. Children living in rural areas have higher rates of obesity than their urban counterparts. Based upon our extensive prior work, the investigators propose a multilevel factorial design randomized controlled trial with interventions at the clinic and individual patient level to treat pediatric obesity among underserved rural children and families. The individual intervention is an mHealth rurally tailored pediatric obesity behavioral intervention (iAmHealthy) vs. Newsletter control while the clinic level intervention is a cluster randomized stepped wedge (Healthy Clinic intervention) designed to improve clinics' treatment of children with overweight and obesity. The iAmHealthy intervention is a rurally tailored empirically supported family-based behavioral group program targeting the families of children who are overweight or obese and providing 26 contact hours of group and individual intervention. The Healthy Clinic intervention is designed to improve provider office processes using a bundled intervention of provider prompts, skills training and intervention tools implemented with performance feedback targeted at the implementation of the American Academy of Pediatrics 2023 Clinical Practice Guideline. This study will be the first to assess both clinic level and patient level pediatric obesity interventions tailored to the unique barriers in rural pediatric populations. Four states (KS, NE, OK, SC), who are members of the ECHO IDeA State Pediatric Clinical Trials Network (ISPCTN) and participated in a previous feasibility study of the iAmHealthy intervention (NCT04142034) in rural medical clinics have each recruited four medical clinics who care for rural children. In each rural clinic, investigators will recruit up to 64 caregiver/child dyads who will be randomly assigned to iAmHealthy or Newsletter, for a total of 512 child/caregiver dyads. The current proposal studies two easily disseminable multilevel interventions and their combination to address modifiable risk factors for cancer in rural populations, specifically pediatric obesity. These findings could significantly change the way medical clinics care for the 41% of rural children who are overweight or obese.

ELIGIBILITY:
Inclusion criteria for individual participants:

* Child is ages 6-11 years at consent
* Child BMI %ile is ≥85th
* Child lives in a rural area
* Child/family speaks English or Spanish

Exclusion criteria for individual participants:

* Child has a physical limitation or injury that substantially limits physical mobility or has a planned medical treatment during the course of the trial that will substantially limit physical mobility
* Child has a known medical issue that could affect protocol compliance (e.g., cancer)
* Child and/or primary caregiver has a developmental delay or cognitive impairment that could affect protocol compliance
* Child is enrolled in a weight-loss trial
* Child has a sibling who has already consented in the trial

Inclusion criteria for clinics:

* History of collaboration with site awardee in research or quality improvement projects
* In the past year at least 300 eligible potential participants
* The clinic must have an electronic medical records system

Exclusion criteria for clinics:

* Unable to generate lists of children seen in clinic by date of visit, age, and zip code

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1024 (Estimated)
Dates: Start 2025-09-06 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 6 months to year 4 in child body mass index (BMI) | Baseline, 6 months, year 4
  Height and weight will be collected remotely and used to calculate BMI, BMIz, BMI%ile and BMI%95th%ile.
Clinic: Independent clinic chart audit | Every six months for 3.5 years
  The primary outcome measure for the Healthy Clinics intervention will be a random audit of 40 medical records in each clinic every 6 months performed by highly trained research staff in each state who are fully independent of the participating medical clinic. The medical record, index visit and latest well visit (within that 6 months), will be audited for child BMI and BMI%ile, evidence of recognition of whether the patient has overweight/obesity, plan for addressing overweight/obesity, followup plan, and counseling for diet and activity. The purpose of the clinic chart audit is to assess the clinic's current activities around identification and treatment of overweight and obesity.

SECONDARY OUTCOMES:
Change from baseline to 6 months to year 4 in child physical activity using the Exercise Vital Sign | Baseline, 6 months, year 4
  The Exercise Vital Sign (EVS) is a modification of the Behavioral Risk Factor Surveillance System (BRFSS) Physical Activity (PA) questions, and its development was supported by PA experts as part of the Exercise is Medicine effort in the United States. EVS assesses the average time spent exercising by multiplying responses on 2 self-reported questions. Responses are multiplied to display minutes per day of moderate or strenuous exercise.
Change from baseline to 6 months to year 4 in child physical activity using the "moderate to vigorous physical activity" screening measure | Baseline, 6 months, year 4
  The "moderate to vigorous physical activity" screening measure is a 2-item parent reported measure.
Change from baseline to 6 months to year 4 in child physical activity using the PROMIS Parent Proxy Physical Activity Measure | Baseline, 6 months, year 4
  The PROMIS Parent Proxy Physical Activity Measure will measure how often parents report in the past 7 days that their child engaged in various physical activity.
Change from baseline to 6 months to year 4 in child dietary behavior | Baseline, 6 months, year 4
  Child dietary behavior will be assessed with the Children's Eating Habits Questionnaire food frequency section (CEHQ-FFQ). The CEHQ-FFQ was designed to estimate the eating behaviors and intakes for each of the major food groups related to general health status and childhood obesity. A conversion factor is used to transform child dietary intake and fast-food consumption into weekly consumption frequencies, ranging from 0 to 25 and 0 to 8, respectively.
Change from baseline to 6 months to year 4 in child sleep | Baseline, 6 months, year 4
  Child sleep will be assessed with the Children's Sleep Habits Questionnaire (CSHQ). This 22-item questionnaire has 9 questions about bedtime, 7 questions about sleep behavior, 2 questions about waking at night, and 4 questions about morning wake up. The measure results in a score of overall sleep quality, with scores over 41 indicating sleep problems.
Parent and child satisfaction of intervention and technology | 6 months
  The child satisfaction measure was developed specifically for the current study and will shadow the parent satisfaction items. Specific to technology, the investigators will also administer the 12-item Parent-Reported Satisfaction Measure, assessing three technology-related satisfaction domains: technical, comfort with technology and perceived privacy, and access.
Change from baseline to 6 months to year 4 in caregiver body mass index (BMI) | Baseline, 6 months, year 4
  Height and weight will be collected remotely and used to calculate BMI.
Clinic: Internal clinic chart audit | Every month for 6 months
  As a measure of interim progress in the Healthy Clinic intervention, clinic staff will conduct monthly audits of their own patient medical records for child BMI and BMI%ile, evidence of recognition of whether the patient has overweight/obesity, plan for addressing overweight/obesity, and counseling for diet and activity. Each audit will include 10 of the most recently seen patients 6-11 years of age who have overweight or obesity. Additional items will be added to assess the individual clinics' ongoing QI process. This will occur only while clinics are in the Healthy Clinics Intervention.

OTHER OUTCOMES:
Child/caregiver demographics and medical history/update | Baseline, 6 months, year 4
  Age, race, ethnicity, income, insurance type (public/private), individuals living in the home, comorbidity conditions, rurality.
Clinic: Qualitative interviews | Year 4
  Study team will conduct structured interviews with participating clinic staff to assess a series of structured questions regarding the barriers and facilitators of: 1. the Healthy Clinic intervention; 2. The iAmHealthy/Newsletter intervention; 3. other aspects of the study including measurement and communication. These interviews will be transcribed and analyzed using the accepted qualitative analysis techniques of Morgan and Krueger.
Clinic: Questionnaires for quality improvement | Years 1 and 4
  Questionnaires will collect quality improvement experience.
Clinic: Questionnaires for current policies/procedures | Years 1 and 4
  Questionnaires will collect current policies/procedures related to overweight and obesity.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Davis, PhD, MPH, ABPP, Principal Investigator — University of Kansas Medical Center; Paul M Darden, MD, Principal Investigator — The University Of Oklahoma Health Sciences Center
Locations (4):
- United States (4):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No